CLINICAL TRIAL: NCT05900882
Title: An Open Label, Single Arm, Multi-Center Exploratory Study to Evaluate the Efficacy and Safety of SVRd for the Treatment of Newly Diagnosed Multiple Myeloma Patients Presenting With Extramedullary Disease.
Brief Title: SVRd for the Treatment of Newly Diagnosed Multiple Myeloma Patients Presenting With Extramedullary Disease
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SVRd
Record Dates: First submitted 2023-05-29; First posted 2023-06-13 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2024-08

CONDITIONS: Multiple Myeloma
Keywords: NDMM; Extramedullary disease; SVRd
MeSH Terms: conditions — Multiple Myeloma | interventions — selinexor; Bortezomib; Lenalidomide; Dexamethasone; Fumigant 93

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- study group (Experimental): SVRd induction treatment
  Interventions: Drug: Selinexor; Drug: Bortezomib; Drug: Lenalidomide; Drug: Dexamethasone

INTERVENTIONS:
Drug: Selinexor — Selinexor 60 mg/day, orally on d1,8,15,22
  Other Names: S
Drug: Bortezomib — Bortezomib 1.3mg/m2 intravenously on d1,8,15,22
  Other Names: V
Drug: Lenalidomide — Lenalidomide 25 mg/d (the dose will be adjusted according to creatinine clearance)
  Other Names: R
Drug: Dexamethasone — Dexamethasone 20 mg/day orally on d1-2, d8-9,d15-16,d22-23
  Other Names: d

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of SVRd in NDMM patients presenting with extramedullary disease.

DETAILED DESCRIPTION:
Study Design:

This protocol corresponds to a multicenter, open-label, single arm, exploratory study designed to determine the safety of the combination of selinexor combined with VRd in NDMM patients presenting with EMD. The patients who respond to this combination treatment will undergo allogeneic hematopoietic stem cell transplantation or no ASCT and followed by consolidation and maintenance treatment.

All patients will receive 4 courses of SVRd induction therapy, each cycle of treatment will compromise 4 weeks of Selinexor 60mg QW treatment. Transplantation could be performed after 2 courses of VRd consolidation therapy. If not receive transplantation will give 4 cycles of SVRd consolidation therapy. Maintenance treatment will continued for a maximum of 2 years.

Study design allows 35 patients. Induction treatment will consist of Selinexor 60 mg/day orally on d1,8,15,22, Bortezomib 1.3mg/m2 intravenously on d1,8,15,22, Lenalidomide 25 mg/d ( the dose will be adjusted according to creatinine clearance), orally on days 1 to14, Dexamethasone 20 mg/day orally on d1-2, d8-9,d15-16,d22-23

ELIGIBILITY:
Inclusion Criteria:

1. Men and women aged with18-75 years old.
2. Confirmed diagnosis of Multiple Myeloma(MM) (IMWG consensus guidelines)
3. Newly diagnosed patients presenting with extramedullary disease (EMD) including solely paraskeletal plasmacytoma, plasmacytoma of soft tissue and other special sites detected by physical exam and confirmed by CT/MRI/PET-CT and/or biopsy (≥2cm).
4. ANC≥1.0*10^9/L, HGB≥75*10^9/L, PLT≥50*10^9/L (≥50% of bone marrow nucleated cells are plasma cells).
5. Patients whose expecting survival time will be more than 3 months.
6. Without active infectious disease.
7. Female patients of child-bearing potential must have a negative serum pregnancy test at screening and all patients agree to use two reliable methods of contraception for six months after their last dose of medication.
8. Willingness and ability to comply with scheduled visits, treatment plans, laboratory tests and other study procedures.
9. Each patient must sign an informed consent form (ICF) indicating that he or she understands the purpose of and procedures required for the study and are willing to participate in the study.

Exclusion Criteria:

1. Patients who have HBV, HCV, and other acquired and congenital immunodeficiency diseases.
2. Patients who have grade 2 or higher of peripheral neuropathy or neuralgia according to the definition of NCI CTCAE version 4.0.
3. Plasma cell leukemia.
4. Serious thrombotic events.
5. Active, unstable cardiovascular dysfunction: a. symptomatic ischemia; b. Uncontrolled, clinically significant conduction abnormalities (except antiarrhythmic ventricular tachycardia), but patients with first-degree atrioventricular block or asymptomatic left anterior bundle/right fascicular block cannot be excluded. c. New York Heart Association (NYHA) Class III - IV or left ventricular ejection fraction (LVEF) <40%; d. Myocardial infarction Within 3 months before C1D1.
6. Significant hepatic dysfunction (ALT and AST ≥ 3 times the upper limit of normal (ULN)).
7. Serum bilirubin≥1.5 × ULN.
8. creatinine clearance <30 ml/min.
9. History of active malignancy during the past 5 years with the exception of basal carcinoma of the skin or stage 0 cervical carcinoma.
10. Previous major operation within 30 days before C1D1.
11. Patients who have epilepsy, dementia requiring medication, or other mental disorders who are unable to understand or adhere to the study protocol.
12. According to the study protocol or in the opinion of the investigator,serious physical or mental illness that is likely to interfere with the study procedures/results.
13. Any psychological, familial, sociological and geographical condition potentially hampering compliance with the study protocol and follow-up schedule.
14. Current participation in another clinical trial.
15. Pregnant or lactating women.
16. Patients with other commodities that the investigators considered not suitable for the enrollment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2022-07-15 (Actual); Primary Completion 2025-08-30 (Estimated); Study Completion 2025-08-30 (Estimated)

PRIMARY OUTCOMES:
Number of Participants With Overall Response Rate (ORR) | End of induction treatment (4 cycles, each cycle is 28 days)
  ORR: defined as the proportion of patients who will achieve PR or better, as per IMWG criteria.

SECONDARY OUTCOMES:
Number of Participants With Complete Response Rate (CR) | End of induction treatment (4 cycles, each cycle is 28 days)
  CR: defined as the proportion of patients who will achieve CR, as per IMWG criteria.
Duration of Response (DOR) | 5 years
  DOR: defined as time, in months, from initial response (PR or better) until the date of a disease progression event
Progression-Free Survival (PFS) | 5 years
  PFS: was calculated from the time of informed consent to the date of recurrence or death, whichever occurred first. Patients were censored at the date of the last follow-up visit if they were alive without relapse.
Overall Survival (OS) | 5 years
  OS was calculated from the date of informed consent to the date of death. Patients still alive at the end of follow-up were censored at the last date of follow-up.
Number of adverse events | During of induction treatment (4 cycles, each cycle is 28 days)
  Adverse events are evaluated with CTCAE V5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Lijuan Chen, Study Chair — The First Affiliated Hospital with Nanjing Medical University
Locations (6):
- China (6):
  - Changzhou Second People's Hospital, Changzhou, Jiangsu
  - Nanjing First People's Hospital, Nanjing, Jiangsu
  - The First Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu
  - Affiliated Hospital of Nantong University, Nantong, Jiangsu
  - Taizhou People's Hospital, Taizhou, Jiangsu
  - Yancheng First People's Hospital, Yancheng, Jiangsu

REFERENCES:
- [Derived] Jin Y, Cheng X, Zhang X, Shi Q, Zhu Y, Li J, Fan L, Chen L. Efficacy and Safety of Selinexor Combined with VRD in Newly Diagnosed Multiple Myeloma with EMD: A Phase 2 Trial. Blood Adv. 2026 Jan 21:bloodadvances.2025018945. doi: 10.1182/bloodadvances.2025018945. Online ahead of print. PMID 41564431